CLINICAL TRIAL: NCT01657305
Title: Open, Blindly Evaluated, Prospective, Controlled, Randomized, Multicenter Phase III Clinical Trial to Compare Intra-individually the Efficacy and Tolerance of Oleogel-S10 Versus Standard of Care in Accelerating the Wound Healing of Split-Thickness Skin Graft Donor Sites
Brief Title: Oleogel-S10 in Wound Healing of Split-Thickness Skin Graft Donor Sites (BSH-12)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Birken AG (Industry)
Responsible Party: Sponsor
Organization: Amryt Pharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BSH-12; 2012-000777-23 (EudraCT Number)
Record Dates: First submitted 2012-07-29; First posted 2012-08-06 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-05

CONDITIONS: Wounds
Keywords: Split-Thickness Skin Graft (STSG) donor site; Split-thickness skin graft; STSG; Wound healing; Skin grafting; Superficial wound; Partial-thickness wound; Time to wound closure
MeSH Terms: conditions — Wounds and Injuries | interventions — episalvan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oleogel-S10, non-adhesive wound dressing (Experimental): A split-thickness skin graft (STSG) donor site wound >15cm2 in size was divided in 2 halves. One half was randomized to Oleogel-S10 treatment and non-adhesive wound dressing (intra-individual comparison). Oleogel-S10 was administered (1 cm or 100 mg per cm2 wound area corresponding to thickness of about 1 mm or 0.04 inch) every 3 to 4 days until 95% epithelialization of the wound or end of treatment at Day 28.
  Interventions: Drug: Oleogel-S10, non-adhesive wound dressing
- Non-adhesive wound dressing only (Other): A STSG donor site wound >15cm2 in size was divided in 2 halves. One half was randomized to treatment with non-adhesive wound dressing only (intra-individual comparison). Non-adhesive wound dressings are standard of care (SOC) in the treatment of STSG donor sites. Wound dressings were changed every 3 to 4 days until 95% epithelialization of the wound or end of treatment at Day 28.
  Interventions: Device: Non-adhesive wound dressing only

INTERVENTIONS:
Drug: Oleogel-S10, non-adhesive wound dressing — 1 cm or 100 mg Oleogel-S10 per cm2 wound area (corresponds to thickness of approximately 1 mm or 0.04 inch) every 3 to 4 days until 95% epithelialization of the wound or end of treatment at Day 28.
  Other Names: Episalvan®
  Arms: Oleogel-S10, non-adhesive wound dressing
Device: Non-adhesive wound dressing only — Soft silicone faced polyurethane foam dressing such as Mepilex® only every 3 to 4 days until 95% epithelialization of the wound or end of treatment at Day 28.
  Other Names: Mepilex®
  Arms: Non-adhesive wound dressing only

SUMMARY:
The main purpose of this phase III clinical trial was to compare intra-individually the efficacy, safety and tolerability of Oleogel-S10 and non-adhesive wound dressing versus non-adhesive wound dressing only in accelerating the wound healing of Split-Thickness Skin Graft (STSG) donor sites.

DETAILED DESCRIPTION:
Oleogel-S10 has shown efficacy and was well tolerated in previous clinical trials in participants with skin lesions. Especially the results in a previous study with STSG donor sites suggested that Oleogel-S10 should be efficacious and safe in the treatment of superficial wounds.

The present phase III clinical trial in STSG donor sites was initiated to demonstrate wound healing progress, i.e., the time to healing and the grade of epithelialization of the wound.

In this study, STSG donor sites were separated into 2 wound halves. Randomly assigned, 1 wound half was treated with Oleogel-S10 and non-adhesive wound dressing, the other wound half with non-adhesive wound dressing only (standard of care).

Wound healing progress was documented by photos which were assessed by expert reviewers blind to the treatment of the wound halves.

ELIGIBILITY:
Inclusion Criteria:

* Presenting a split-thickness skin graft donor site wound with a minimum size of 15 cm2 and with a minimum width of 3 cm.
* Patient is able to understand the Informed Consent Form (ICF) provided and is prepared to comply with all study requirements, including the following: Visiting the trial site for wound dressing change and photo documentation every third or fourth day until both wound halves are closed (but no longer than 28 days after surgery).
* Willing to perform all necessary wound dressing changes at the trial site. Also the patient needs to agree to return to site for 3 and 12 months follow-up visits.
* Women of childbearing potential must apply highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly (e.g., implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices (IUDs), sexual abstinence, or a vasectomized partner)).

Exclusion Criteria:

* Diseases or conditions that could, in the opinion of the Investigator, interfere with the assessment of safety or efficacy.
* A skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
* A history of clinically significant hypersensitivity to any of the drugs, surgical dressings or excipients to be used in this trial.
* Known multiple allergic disorders.
* Taking, or have taken, any investigational drugs within 3 months prior to the screening visit.
* Pregnant or breast feeding women are not allowed to participate in the study.
* Inappropriate to participate in the study, for any reason, in the opinion of the investigator.
* Mental incapacity or language barriers precluding adequate understanding the Informed consent form or co-operation or willingness to follow study procedures.
* Previous participation in this study.
* Employee at the investigational site, relative or spouse of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Robert Metelmann, Prof, Principal Investigator — Universitätsmedizin Greifswald MKG-Chirurgie/Plastische Operationen
Locations (24):
- Austria (3):
  - Medical University of Graz, Graz
  - Landesklinik für Dermatologie, Salzburg
  - Medical University Vienna, Vienna
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment-"Dr. Georgi Stranski" EAD, Pleven
  - University Multiprofile Hospital for Active Treatment "Saint George", Plovdiv
  - Multiprofile Hospital for Active Treatment- Ruse, Rousse
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine "N.I.Pirogov", Sofia
  - University Multiprofile Hospital for Active Treatment-Varna at MMA-Sofia, Varna
- Czechia (2):
  - Universtity Hospital Brno, Brno
  - University Hospital Olomouc, Olomouc
- Finland (2):
  - Päijät-Hämeen keskussairaala, Lahti
  - Satakunnan keskussairaala, Pori
- Germany (10):
  - Trauma Hospital, Berlin
  - University Hospital, Düsseldorf
  - Essen University Hospital, Essen
  - University Hospital, Frankfurt
  - University Medical Center, Freiburg im Breisgau
  - University Medicine Greifswald, Greifswald
  - HELIOS Clinic, Krefeld
  - University Medical Center, Mainz
  - Klinikum rechts der Isar, München
  - Klinikum Offenbach am Main, Offenbach
- Poland (2):
  - Univesity Hospital Gdansk, Gdansk
  - Samodzelny Publiczny Szpital Kliniczny Nr. 1, Lublin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barret JP, Podmelle F, Lipovy B, Rennekampff HO, Schumann H, Schwieger-Briel A, Zahn TR, Metelmann HR; BSH-12 and BSG-12 study groups. Accelerated re-epithelialization of partial-thickness skin wounds by a topical betulin gel: Results of a randomized phase III clinical trials program. Burns. 2017 Sep;43(6):1284-1294. doi: 10.1016/j.burns.2017.03.005. Epub 2017 Apr 8. PMID 28400148

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 03 Aug 2012 to 01 Aug 2013 in 18 clinical centers in 6 countries: Germany (8 centers), Czech Republic (2 centers), Poland (1 center), Finland (1 center), Austria (2 centers), and Bulgaria (4 centers).
Pre-assignment Details: 111 participants were screened and wound halves of 107 participants were randomized and treated. For four screened participants, wound halves were neither randomized nor treated with study medication for the following reasons: not randomized by mistake, violation of inclusion criteria, surgery cancelled, and withdrawal of consent.
Groups:
- Entire Study Population: Intraindividual comparison: A split-thickness skin graft (STSG) donor site wound ≥15 cm² in size was divided in 2 halves. One wound half was randomized to Oleogel-S10 treatment and non-adhesive wound dressing, the other half to non-adhesive wound dressing (intra-individual comparison). Non-adhesive wound dressings such as soft silicone-faced polyurethane foam dressings (e.g., Mepilex®) represent standard of care (SOC) in the treatment of STSG donor site wounds. Oleogel-S10 was administered at a thickness of approximately 1 mm or 0.04 inches. Treatment was repeated and wound dressings were changed at least every 3 to 4 days until wound closure (at least 95% epithelialisation) was achieved or the end of treatment was reached at Day 28.
Period: Overall Study
Arm/Group | Entire Study Population
Started | 107
Completed | 82
Not Completed | 25
Not completed — Lack of Wound Closure at Day 28 | 15
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Did not Adhere to Protocol/Procedures | 4

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Intra-individual comparison: A split-thickness skin graft (STSG) donor site wound ≥15 cm² in size was divided in 2 halves. One half was randomized to Oleogel-S10 treatment and non-adhesive wound dressing, the other half to non-adhesive wound dressing only. Non-adhesive wound dressings, specifically soft silicone faced polyurethane foam dressings (e.g., Mepilex®), represent standard of care (SOC) in the treatment of STSG donor site wounds. Oleogel-S10 was administered at a thickness of 1 mm (0.04 inches) and wound dressings were changed at least every 3 to 4 days. Study treatment continued until both wound halves were closed (at least 95% epithelialised) or ended at Day 28.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 65
  >=65 years | 40
Age, Continuous [Median (Full Range); unit: years] | 56 [18 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 68
Region of Enrollment [Number; unit: participants]
  Czech Republic | 40
  Austria | 4
  Finland | 3
  Poland | 2
  Bulgaria | 24
  Germany | 34

OUTCOME MEASURES:

1. Primary Outcome: Intra-individual Difference in Time to Wound Closure
Description: Intra-individual difference in time to wound closure between wound halves, either treated with Oleogel-S10 and non-adhesive wound dressing or treated with non-adhesive wound dressing only. Independent experts were blind to treatment and assessed efficacy based on chronological series of cropped and coded photographs by wound half that were taken before start of treatment, during wound dressing changes and at the end of treatment. Difference in time to wound closure was calculated for every individual participant as [time taken for wound half treated with Oleogel-S10 to close] - [time taken for wound half treated with non-adhesive wound dressing to close], i.e., results below 0 indicate earlier wound closure of Oleogel-S10 treatment. The overall mean difference in time to wound closure was calculated based on all mean differences in time to wound closure of individual participants. Hence, primary outcome data derived from mean difference in time to wound closure by participant.
Time Frame: up to 4 weeks
Population: The intent-to-treat (ITT) analysis population included all participants who were treated at least once with study medication, i.e. who received any dose of Oleogel-S10.
Measure: Mean (95% Confidence Interval); unit: days
Groups:
- Entire Study Population: All patients treated with Oleogel-S10 plus non-adhesive wound dressing and with non-adhesive wound dressing only.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 107
days | -1.4 [-1.8 to -0.9]
Statistical Analysis 1: Comparison: Entire Study Population; All participants received both treatments and treatments were intra-individually compared. Hypotheses tested: H0: δ = 0 and H1: δ ≠ 0 with δ being the difference in time to wound closure between treatments. Negative values for the intra-individual time difference indicate faster healing of the Oleogel-S10-treated wound half. For right-censored observations (no wound closure observed in blinded photo evaluation), wound closure was conservatively calculated as +1 day after the last photo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — 2-sided, significance level = 0.05

2. Secondary Outcome: Time From Surgery Until Wound Closure is Achieved
Description: Time from surgery until wound closure is achieved, separately for wound halves treated with Oleogel-S10 and non-adhesive wound dressing vs. non-adhesive wound dressing only. While outcome measure 1 (intra-individual difference in time to wound closure) was calculated based on mean intra-individual difference in time to wound closure in 107 participants with missing values replaced by a value of 0, for outcome measure 2 missing values were not replaced. For 5 of the 107 wounds data were missing, thus the reported values are calculated from 102 STSG donor site wound halves by intervention (Oleogel-S10 and non-adhesive wound dressing vs. non-adhesive wound dressing only).
Time Frame: up to 4 weeks
Population: The intent-to-treat (ITT) analysis population included all participants who were treated at least once with study medication, i.e. who received any dose of Oleogel-S10 and who had signed an informed consent form. For 5 of the 107 wounds, data were missing, thus the reported values are calculated from 102 STSG donor site wound halves by intervention
Measure: Mean (95% Confidence Interval); unit: Days from surgery until wound closure
Units Other Than Participants: Number of STSG wound (halves) analyzed
Groups:
- Oleogel-S10, Non-adhesive Wound Dressing: A split-thickness skin graft (STSG) donor site wound >15cm2 in size was divided in 2 halves. One half was randomized to Oleogel-S10 treatment and non-adhesive wound dressing (intra-individual comparison). Oleogel-S10 was administered (1 cm or 100 mg per cm2 wound area corresponding to thickness of about 1 mm or 0.04 inches) every 3 to 4 days until 95% epithelialization of the wound or end of treatment at Day 28.
  Oleogel-S10, non-adhesive wound dressing: 1 cm or 100 mg Oleogel-S10 per cm2 wound area (corresponds to thickness of approximately 1 mm or 0.04 inches) every 3 to 4 days until 95% epithelialization of the wound or end of treatment at Day 28.
Arm/Group | Oleogel-S10, Non-adhesive Wound Dressing | Non-adhesive Wound Dressing Only
Number analyzed (Participants) | 107 | 107
Number analyzed (Number of STSG wound (halves) analyzed) | 102 | 102
Days from surgery until wound closure | 15.5 [14.2 to 16.8] | 17.1 [15.8 to 18.5]

3. Secondary Outcome: Percentage of Participants With Earlier Healing
Description: Percentage of participants with earlier healing of wound area treated with Oleogel-S10 and non-adhesive wound dressing compared to non-adhesive wound dressing only
Time Frame: up to 4 weeks
Population: The intent-to-treat (ITT) analysis population included all participants who were treated at least once with study medication, i.e. who received any dose of Oleogel-S10 and who had signed an informed consent form.
Measure: Number (95% Confidence Interval); unit: Percentage with earlier healing
Arm/Group | Oleogel-S10, Non-adhesive Wound Dressing | Non-adhesive Wound Dressing Only
Number analyzed (Participants) | 107 | 107
Percentage with earlier healing | 61.7 [51.8 to 70.9] | 7.5 [3.3 to 14.2]

4. Secondary Outcome: Percentage of Participants With Wound Closure at Different Time Points
Description: For separate time points (Day 7, Day 10, Day 14, Day 18, Day 21, and Day 28), the frequencies of wound areas which have reached wound closure were calculated.
Time Frame: up to 4 weeks
Population: The intent-to-treat (ITT) analysis population included all participants who were treated at least once with study medication, i.e. who received any dose of Oleogel-S10 and who had signed an informed consent form. Data were missing for n=5 participants at all time points.
Measure: Number (95% Confidence Interval); unit: Percentage with wound closure
Arm/Group | Oleogel-S10, Non-adhesive Wound Dressing | Non-adhesive Wound Dressing Only
Number analyzed (Participants) | 102 | 102
Percentage with wound closure
  Day 7 | 2.0 [0.2 to 6.9] | 1.0 [0.0 to 5.3]
  Day 10 | 25.5 [17.4 to 35.1] | 15.7 [9.2 to 24.2]
  Day 14 | 49.0 [39.0 to 59.1] | 37.3 [27.9 to 47.4]
  Day 18 | 70.6 [60.7 to 79.2] | 61.8 [51.6 to 71.2]
  Day 21 | 77.5 [68.1 to 85.1] | 71.6 [61.8 to 80.1]
  Day 28 | 94.1 [87.6 to 97.8] | 90.2 [82.7 to 95.2]

5. Secondary Outcome: Percentage of Wound Epithelialization at Different Time Points as Assessed by the Investigator
Description: A study team member assessed the progress of wound healing by treatment regimen and noted the degree of epithelialization (expressed in percent of the original wound size) at wound dressing changes on Day 7, Day 10, Day 14, Day 18, Day 21, and Day 28.
Time Frame: up to 4 weeks
Population: The intent-to-treat (ITT) analysis population included all participants who were treated at least once with study medication, i.e. who received any dose of Oleogel-S10 and who had signed an informed consent form. Data were missing for n=1 participant at all time points.
Measure: Mean (95% Confidence Interval); unit: Area Percent of initial wound size
Arm/Group | Oleogel-S10, Non-adhesive Wound Dressing | Non-adhesive Wound Dressing Only
Number analyzed (Participants) | 107 | 107
Area Percent of initial wound size
  Day 7: number analyzed (Participants) | 106 | 106
  Day 7 | 36.7 [30.4 to 43.0] | 28.1 [22.3 to 33.9]
  Day 10: number analyzed (Participants) | 106 | 106
  Day 10 | 60.0 [52.9 to 67.1] | 49.9 [43.0 to 56.7]
  Day 14: number analyzed (Participants) | 106 | 106
  Day 14 | 82.2 [76.9 to 87.5] | 74.3 [68.5 to 80.1]
  Day 18: number analyzed (Participants) | 106 | 106
  Day 18 | 89.7 [85.4 to 93.9] | 82.3 [77.3 to 87.3]
  Day 21: number analyzed (Participants) | 106 | 106
  Day 21 | 92.2 [88.6 to 95.9] | 85.8 [81.3 to 90.4]
  Day 28: number analyzed (Participants) | 106 | 106
  Day 28 | 93.9 [90.6 to 97.2] | 90.0 [85.9 to 94.0]
Statistical Analysis 1: Comparison: Oleogel-S10, Non-adhesive Wound Dressing vs Non-adhesive Wound Dressing Only; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Day 7; Mean Difference (Final Values) = 8.6, 95% CI 2-sided [6.0 to 11.2], Standard Deviation 13.4 — Difference in degree of epithelialization [%] (Oleogel-S10 minus standard of care)
Statistical Analysis 2: Comparison: Oleogel-S10, Non-adhesive Wound Dressing vs Non-adhesive Wound Dressing Only; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Day 10; Mean Difference (Final Values) = 10.1, 95% CI 2-sided [6.9 to 13.4], Standard Deviation 17.0 — Difference in degree of epithelialization [%] (Oleogel-S10 minus standard of care)
Statistical Analysis 3: Comparison: Oleogel-S10, Non-adhesive Wound Dressing vs Non-adhesive Wound Dressing Only; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Day 14; Mean Difference (Final Values) = 7.9, 95% CI 2-sided [4.6 to 11.1], Standard Deviation 17.0 — Difference in degree of epithelialization [%] (Oleogel-S10 minus standard of care)
Statistical Analysis 4: Comparison: Oleogel-S10, Non-adhesive Wound Dressing vs Non-adhesive Wound Dressing Only; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Day 18; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [3.9 to 10.9], Standard Deviation 18.3 — Difference in degree of epithelialization [%] (Oleogel-S10 minus standard of care)
Statistical Analysis 5: Comparison: Oleogel-S10, Non-adhesive Wound Dressing vs Non-adhesive Wound Dressing Only; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Day 21; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [3.7 to 9.1], Standard Deviation 14.1 — Difference in degree of epithelialization [%] (Oleogel-S10 minus standard of care)
Statistical Analysis 6: Comparison: Oleogel-S10, Non-adhesive Wound Dressing vs Non-adhesive Wound Dressing Only; Test type: Superiority or Other; p = 0.0021, t-test, 2 sided — Day 28; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [1.5 to 6.4], Standard Deviation 12.9 — Difference in degree of epithelialization [%] (Oleogel-S10 minus standard of care)

6. Secondary Outcome: Likert Scale Rating of Efficacy
Description: Participants and investigators were asked to grade the efficacy of Oleogel-S10 and non-adhesive wound dressing versus non-adhesive wound dressing only on a 5-point Likert scale (treatment with Oleogel-S10 is much more effective, treatment with Oleogel-S10 is more effective, both treatments have the same efficacy, non-adhesive wound dressing only is more effective, non-adhesive wound dressing only is much more effective).
Time Frame: up to 4 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of efficacy asssessments
Groups:
- Investigator Asssessment Day 7: Efficacy as assessed by investigator at Day 7
- Investigator Assessment Day 14: Efficacy as assessed by investigator at Day 14
- Investigator Assessment Day 21: Efficacy as assessed by investigator at Day 21
- Investigator Assessment Day 28: Efficacy as assessed by investigator at Day 28
- Investigator Assessment End of Treatment: Efficacy as assessed by investigator at End of Treatment (EoT)
- Participant Assessment Day 7: Efficacy as assessed by participant at Day 7
- Participant Assessment Day 14: Efficacy as assessed by participant at Day 14
- Participant Assessment Day 21: Efficacy as assessed by participant at Day 21
- Participant Assessment Day 28: Efficacy as assessed by participant at Day 28
- Participant Assessment EoT: Efficacy as assessed by participant at EoT
Arm/Group | Investigator Asssessment Day 7 | Investigator Assessment Day 14 | Investigator Assessment Day 21 | Investigator Assessment Day 28 | Investigator Assessment End of Treatment | Participant Assessment Day 7 | Participant Assessment Day 14 | Participant Assessment Day 21 | Participant Assessment Day 28 | Participant Assessment EoT
Number analyzed (Participants) | 100 | 101 | 97 | 95 | 104 | 100 | 101 | 97 | 95 | 104
Percentage of efficacy asssessments
  Oleogel-S10 much more effective | 15.0 [8.6 to 23.5] | 20.8 [13.4 to 30.0] | 19.6 [12.2 to 28.9] | 15.8 [9.1 to 24.7] | 16.3 [9.8 to 24.9] | 18.0 [11.0 to 26.9] | 15.8 [9.3 to 24.4] | 21.6 [13.9 to 31.2] | 20.0 [12.5 to 29.5] | 21.2 [13.8 to 30.3]
  Oleogel-S10 more effective | 46.0 [36.0 to 56.3] | 49.5 [39.4 to 59.6] | 51.5 [41.2 to 61.8] | 52.6 [42.1 to 63.0] | 51.9 [41.9 to 61.8] | 44.0 [34.1 to 54.3] | 46.5 [36.5 to 56.7] | 42.3 [32.3 to 52.7] | 42.1 [32.0 to 52.7] | 41.3 [31.8 to 51.4]
  Both treatments same efficacy | 31.0 [22.1 to 41.0] | 24.8 [16.7 to 34.3] | 25.8 [17.4 to 35.7] | 29.5 [20.6 to 39.7] | 28.8 [20.4 to 38.6] | 33.0 [23.9 to 43.1] | 31.7 [22.8 to 41.7] | 32.0 [22.9 to 42.2] | 34.7 [25.3 to 45.2] | 34.6 [25.6 to 44.6]
  Standard of care (SOC) more effective | 8.0 [3.5 to 15.2] | 3.0 [0.6 to 8.4] | 1.0 [0.0 to 5.6] | 1.1 [0.0 to 5.7] | 1.9 [0.2 to 6.8] | 5.0 [1.6 to 11.3] | 4.0 [1.1 to 9.8] | 3.1 [0.6 to 8.8] | 3.2 [0.7 to 9.0] | 2.9 [0.6 to 8.2]
  SOC much more effective | 0.0 [0.0 to 0.0] | 2.0 [0.2 to 7.0] | 2.1 [0.3 to 7.3] | 1.1 [0.0 to 5.7] | 1.0 [0.0 to 5.2] | 0.0 [0.0 to 0.0] | 2.0 [0.2 to 7.0] | 1.0 [0.0 to 5.6] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

7. Secondary Outcome: Cosmetic Outcome at 3 and 12 Months After Surgery, Respectively
Description: Blinded photographic evaluation which wound half resembles more closely the surrounding skin with regard to texture, redness, growth of hair, and pigmentation.
Time Frame: 3 months and 12 months
Population: The intent-to-treat (ITT) analysis population included 87 participants for the 3-months follow-up and 83 participants for the 12-months follow-up.
Measure: Number (95% Confidence Interval); unit: Percentage of wounds
Groups:
- Texture at 3 Months Follow-up: Evaluation of cosmetic outcome with regard to texture at 3 months follow-up
- Hair Growth at 3 Months Follow-up: Evaluation of cosmetic outcome with regard to hair growth at 3 months follow-up
- Pigmentation at 3 Months Follow-up: Evaluation of cosmetic outcome with regard to pigmentation at 3 months follow-up
- Redness at 3 Months Follow-up: Evaluation of cosmetic outcome with regard to redness at 3 months follow-up
- Texture at 12 Months Follow-up: Evaluation of cosmetic outcome with regard to texture at 12 months follow-up
- Hair Growth at 12 Months Follow-up: Evaluation of cosmetic outcome with regard to hair growth at 12 months follow-up
- Pigmentation at 12 Months Follow-up: Evaluation of cosmetic outcome with regard to pigmentation at 12 months follow-up
- Redness at 12 Months Follow-up: Evaluation of cosmetic outcome with regard to redness at 12 months follow-up
Arm/Group | Texture at 3 Months Follow-up | Hair Growth at 3 Months Follow-up | Pigmentation at 3 Months Follow-up | Redness at 3 Months Follow-up | Texture at 12 Months Follow-up | Hair Growth at 12 Months Follow-up | Pigmentation at 12 Months Follow-up | Redness at 12 Months Follow-up
Number analyzed (Participants) | 87 | 87 | 87 | 87 | 83 | 83 | 83 | 83
Percentage of wounds
  Wound half treated with Oleogel-S10 | 36.8 [26.7 to 47.8] | 1.1 [0.0 to 6.2] | 41.4 [30.9 to 52.4] | 31.0 [21.5 to 41.9] | 13.3 [6.8 to 22.5] | 2.4 [0.3 to 8.4] | 20.5 [12.4 to 30.8] | 10.8 [5.1 to 19.6]
  Wound half treated with wound dressing only | 5.7 [1.9 to 12.9] | 0.0 [0.0 to 0.0] | 6.9 [2.6 to 14.4] | 5.7 [1.9 to 12.9] | 2.4 [0.3 to 8.4] | 1.2 [0.0 to 6.5] | 8.4 [3.5 to 16.6] | 3.6 [0.8 to 10.2]
  Both equal | 51.7 [40.8 to 62.6] | 97.7 [91.9 to 99.7] | 47.1 [36.3 to 58.1] | 58.6 [47.6 to 69.1] | 84.3 [74.7 to 91.4] | 96.4 [89.8 to 99.2] | 68.7 [57.6 to 78.4] | 85.5 [76.1 to 92.3]

8. Secondary Outcome: Likert Scale Rating of Tolerability
Description: Participants and investigators were asked to evaluate the tolerability of Oleogel-S10 and non-adhesive wound dressing versus non-adhesive wound dressing only (standard of care) on a 5-point Likert scale (treatment with Oleogel-S10 is much better tolerated, treatment with Oleogel-S10 is better tolerated, both treatments are equally well tolerated, standard of care is better tolerated, standard of care is much better tolerated).
Time Frame: up to 4 weeks
Population: The safety analysis population (SAF) included all participants who received treatment at least once, i.e. who received any dose of Oleogel-S10 or standard of care (SOC). If the application of any treatment was uncertain, the participant was included in the SAF.
Measure: Number; unit: Percentage of participants
Groups:
- Investigator Asssessment Day 7: Tolerability as assessed by investigator at Day 7
- Investigator Assessment Day 14: Tolerability as assessed by investigator at Day 14
- Investigator Assessment Day 21: Tolerability as assessed by investigator at Day 21
- Investigator Assessment Day 28: Tolerability as assessed by investigator at Day 28
- Investigator Assessment End of Treatment: Tolerability as assessed by investigator at End of Treatment (EoT)
- Participant Assessment Day 7: Tolerability as assessed by participant at Day 7
- Participant Assessment Day 14: Tolerability as assessed by participant at Day 14
- Participant Assessment Day 21: Tolerability as assessed by participant at Day 21
- Participant Assessment Day 28: Tolerability as assessed by participant at Day 28
- Participant Assessment EoT: Tolerability as assessed by participant at EoT
Arm/Group | Investigator Asssessment Day 7 | Investigator Assessment Day 14 | Investigator Assessment Day 21 | Investigator Assessment Day 28 | Investigator Assessment End of Treatment | Participant Assessment Day 7 | Participant Assessment Day 14 | Participant Assessment Day 21 | Participant Assessment Day 28 | Participant Assessment EoT
Number analyzed (Participants) | 107 | 107 | 107 | 107 | 107 | 107 | 107 | 107 | 107 | 107
Percentage of participants
  Oleogeogel-S10 much better tolerated | 6.0 | 9.9 | 14.4 | 11.6 | 11.5 | 10.0 | 7.9 | 16.5 | 12.6 | 13.5
  Oleogel-S10 better tolerated | 38.0 | 40.6 | 32.0 | 32.6 | 33.7 | 34.0 | 37.6 | 29.9 | 31.6 | 30.8
  Both treatments equally well tolerated | 52.0 | 49.5 | 51.5 | 55.8 | 54.8 | 53.0 | 50.5 | 51.5 | 54.7 | 54.8
  SOC better tolerated | 4.0 | 0.0 | 2.1 | 0.0 | 0.0 | 3.0 | 4.0 | 2.1 | 1.1 | 1.0
  SOC much better tolerated | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

9. Secondary Outcome: Pharmacokinetic (PK) Data (Number of Plasma Samples With Measurable Betulin Concentration)
Description: Systemic presence/concentration of betulin in blood plasma samples. Plasma samples were collected in weekly intervals and at the end of treatment (when wound closure was achieved or at Day 28). Samples were analysed in a central laboratory with a validated LC-MS/MS method with a lower limit of quantification (LLOQ) of 1 ng/mL.
Time Frame: up to 4 weeks
Population: The safety analysis population included all participants who received treatment at least once, i.e. who received any dose of Oleogel-S10 or standard of care (SOC). If the application of any treatment was uncertain, the participant was included in the SAF.
Measure: Number; unit: Plasma Samples
Units Other Than Participants: Plasma Samples
Groups:
- Day 0 (Pre-dose): Plasma samples collected at the day of STSG surgery prior to first treatment with study medication
- Treatment Period: Plasma samples collected at Day 7, Day 14, Day 21 or at end of treatment (day of wound closure or Day 28)
Arm/Group | Day 0 (Pre-dose) | Treatment Period
Number analyzed (Participants) | 107 | 106
Number analyzed (Plasma Samples) | 107 | 281
Plasma Samples
  Samples below LLOQ (<1 ng/mL) | 105 | 272
  Samples above LLOQ (range in ng/mL) | 2 | 3
  Samples with no valid result | 0 | 6

10. Secondary Outcome: Pharmacokinetic (PK) Data (Plasma Betulin Concentration)
Description: Systemic presence/concentration of betulin in blood plasma samples - values for the number of samples with measurable values in samples above the lower limit of quantification (LLOQ) of 1 ng/mL
Time Frame: up to 4 weeks
Population: A total of 5 participants had a total of 5 samples with betulin concentrations above the LLOQ (1 ng/mL)
Measure: Mean (Full Range); unit: Betulin (ng/mL)
Units Other Than Participants: Samples above LLOQ
Arm/Group | Day 0 (Pre-dose) | Treatment Period
Number analyzed (Participants) | 107 | 106
Number analyzed (Samples above LLOQ) | 2 | 3
Betulin (ng/mL) | 2.1 [1.3 to 3.0] | 2.4 [1.2 to 4.6]

11. Secondary Outcome: Frequency of Adverse Events
Time Frame: Day 0 (start of treatment) until end of treatment (Day 28 or earlier if full wound closure was achieved earlier).
Population: as for outcome 9
Measure: Number; unit: Participants with adverse events (%)
Groups:
- Entire Study Population: All participants who were randomized and treated with Oleogel-S10 and non-adhesive wound dressing and/or non-adhesive wound dressing only.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 107
Participants with adverse events (%)
  Adverse events (AEs) | 17.8
  Serious adverse events | 1.9
  AEs leading to discontinuation | 1.9
  Related AEs | 2.8
  Application site reactions | 8.4

12. Secondary Outcome: Severity of Adverse Events
Description: Adverse Events were graded according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) as being mild (NCI CTCAE Grade 1), moderate (NCI CTCAE Grade 2), severe (NCI CTCAE Grade 3), life-threatening (NCI CTCAE Grade 4) or death (NCI CTCAE Grade 5).
Time Frame: Day 0 (start of treatment) until end of treatment (Day 28 or earlier if full wound closure was achieved earlier).
Population: as for outcome 9
Measure: Number; unit: Participants with adverse events (%)
Arm/Group | Entire Study Population
Number analyzed (Participants) | 107
Participants with adverse events (%)
  Mild (CTCAE Grade 1) | 10.3
  Moderate (CTCAE Grade 2) | 4.7
  Severe (CTCAE Grade 3) | 4.7
  Life-Threatening (CTCAE Grade 4) | 0.0
  Death (CTCAE Grade 5) | 0.0

13. Secondary Outcome: Adverse Events by Relationship to Study Medication
Description: Adverse events were assessed as being 'unlikely', 'possibly' or 'probably' related to study medication, 'not related' to study medication or the relationship to study medication was rated as 'unknown'.
Time Frame: Day 0 (start of treatment) until end of treatment (Day 28 or earlier if full wound closure was achieved earlier).
Population: as for outcome 9
Measure: Number; unit: Participants with adverse events (%)
Arm/Group | Entire Study Population
Number analyzed (Participants) | 107
Participants with adverse events (%)
  'Unlikely' related | 0.0
  'Possibly' related | 2.8
  'Probably' related | 0.0
  Unknown relationship | 0.0
  No relationship | 15.9

ADVERSE EVENTS:
Time Frame: Day 0 (start of treatment) until end of treatment (Day 28 or earlier if full wound closure was achieved earlier).
Groups:
- Entire Study Population - Systemic Adverse Events (AE): All participants treated with Oleogel-S10 plus non-adhesive wound dressing and/or non-adhesive wound dressing only. AEs not localized to any wound application site by the investigator are reported in this arm.
- Oleogel-S10 Localized AE: All participants treated with Oleogel-S10 plus non-adhesive wound dressing and/or non-adhesive wound dressing only. Application site reactions as judged by the investigator which occurred only at the Oleogel-S10 wound half are reported in this arm.
- Non-adhesive Wound Wound Dressing Localized AE: All participants treated with Oleogel-S10 plus non-adhesive wound dressing and/or non-adhesive wound dressing only. Application site reactions as judged by the investigator which occurred only at the wound half treated only with non-adhesive wound dressing are reported in this arm.
- Localized AE Both Wound Halves: All participants treated with Oleogel-S10 plus non-adhesive wound dressing and/or non-adhesive wound dressing only. Application site reactions as judged by the investigator which occurred at both the Oleogel-S10 wound half and the non-adhesive wound dressing only half in one patient are reported in this arm.
Arm/Group | Entire Study Population - Systemic Adverse Events (AE) | Oleogel-S10 Localized AE | Non-adhesive Wound Wound Dressing Localized AE | Localized AE Both Wound Halves
Serious Adverse Events (participants affected / at risk) | 1/107 | 0/107 | 0/107 | 1/107
Other Adverse Events (participants affected / at risk) | 0/107 | 0/107 | 0/107 | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study Population - Systemic Adverse Events (AE) (N=107) | Oleogel-S10 Localized AE (N=107) | Non-adhesive Wound Wound Dressing Localized AE (N=107) | Localized AE Both Wound Halves (N=107)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires approval of the sponsor without specification of an embargo time period.